CLINICAL TRIAL: NCT02355496
Title: The Impact of Charge Displays on Inpatient Laboratory Test Ordering
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 821783
Record Dates: First submitted 2015-01-30; First posted 2015-02-04 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Health Behavior
Keywords: Cost Control; Data Display; Diagnostic Tests, Routine; Physician's Practice Patterns
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Displaying medicare fee data (Experimental): The active arm is the intervention group of randomly selected inpatient laboratory tests (about 15 most frequently ordered and about 15 most expensive) that will have medicare fee data displayed in the computerized provider order entry system.
  Interventions: Other: Displaying medicare fee data
- Control Arm (No Intervention): The control arm is the group of randomly selected inpatient laboratory tests (about 15 most frequently ordered and about 15 most expensive) that will not have medicare fee data displayed.

INTERVENTIONS:
Other: Displaying medicare fee data — Using the computerized order entry system to make medicare fee data for a randomly selected inpatient laboratory tests transparent to providers at the time of order entry.
  Arms: Displaying medicare fee data

SUMMARY:
This is a clinical trial to evaluate the impact of presenting medicare fee data for inpatient laboratory tests in the electronic health record on provider ordering behavior at a tertiary care hospital.

DETAILED DESCRIPTION:
This study is a clinical trial to determine the impact on inpatient laboratory test ordering of presenting providers with medicare fee data at the time of order entry. We will randomly assign 60 laboratory tests to an active arm (medicare fee data displayed) or to a control arm (medicare fee data not displayed). The primary outcome will be the change in the ratio of tests ordered per patient day over 12 months by study group (intervention vs. control).

ELIGIBILITY:
Inclusion Criteria:

* Not applicable

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 98529 (Actual)
Dates: Start 2015-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The ratio of tests ordered per patient-day | 12 months
  Number of tests ordered

SECONDARY OUTCOMES:
The total associated fees of tests ordered per patient-day | 12 months
  Associated costs of test

CONTACTS AND LOCATIONS:
Overall Officials: Mina Sedrak, MD, Study Director — University of Pennsylvania; Mitesh Patel, MD, MBA, MS, Principal Investigator — University of Pennsylvania

REFERENCES:
- [Result] Sedrak MS, Myers JS, Small DS, Nachamkin I, Ziemba JB, Murray D, Kurtzman GW, Zhu J, Wang W, Mincarelli D, Danoski D, Wells BP, Berns JS, Brennan PJ, Hanson CW, Dine CJ, Patel MS. Effect of a Price Transparency Intervention in the Electronic Health Record on Clinician Ordering of Inpatient Laboratory Tests: The PRICE Randomized Clinical Trial. JAMA Intern Med. 2017 Jul 1;177(7):939-945. doi: 10.1001/jamainternmed.2017.1144. PMID 28430829
- See also: Publication in JAMA Internal Medicine — http://jamanetwork.com/journals/jamainternalmedicine/fullarticle/2619519